CLINICAL TRIAL: NCT01785953
Title: CONVENTIONAL AND EXPERIMENTAL CHEMOTHERAPY WITH ALLOGENEIC TRANSPLANT IN YOUNG PATIENTS WITH ACUTE MYELOID LEUKAEMIA
Acronym: AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Benedetto Bruno, MD, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: AML-TO-2012
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is evaluate patients with acute myeloid leukemia (<=66 years), treated with conventional and experimental chemotherapy following allogeneic transplantation. THis patients have been enrolled from 2000 to 2011 at the Division of Hematology, Molinette University Hospital. The purpose of data collection is to assess, with retrospective analysis, the clinical outcome divided by risk class and evaluated in patients who achieve complete remission after induction therapy and consolidation.

ELIGIBILITY:
Patients with acute myeloid leukemia (<=66 years), treated with conventional and experimental chemotherapy following allogeneic transplantation. THis patients have been enrolled from 2000 to 2011 at the Division of Hematology, Molinette University Hospital.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myeloid leukemia patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
Event-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Bruno, MD, Principal Investigator — Divisione di Ematologia-Città della Salute e della Scienza di Torino
Locations (1):
- Città della Salute e della Scienza di Torino, Torino, Italy